CLINICAL TRIAL: NCT01423877
Title: Comparative Effectiveness of Bariatric Surgery Versus Medical Management to Induce Diabetes Remission in Diabetic Patients With BMI 30-35
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-00808
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes
Keywords: bariatric surgery; diabetes; sleeve gastrectomy; gastric bypass; gastric banding
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Specific Aims & Hypothesis Primary Aim: To evaluate laparoscopic bariatric surgery versus intensive medical weight management on indices of insulin resistance and resolution of type 2 diabetes among patients with BMI 30-35.

Hypothesis: Bariatric surgery is the most effective treatment to induce diabetes remission in obese diabetic patients BMI 30-35.

The primary outcomes will be assessed at 6 months: (1) within-patient change in insulin resistance after either bariatric surgery or initiation of intensive medical weight management, and (2) remission of diabetes, (i.e., fasting glucose <126mg/dL and glucose <200mg/dL two hours after a standard 75g oral glucose load without the use of anti-hyperglycemic medications). Insulin resistance will be assessed at randomization and at 6 months with the homeostatic model assessment of insulin resistance (HOMA IR) based on insulin and fasting glucose, as well as oral glucose tolerance tests with area-under-the-curve (AUC) measurement for insulin values. Medication discontinuation will be derived from electronic health records and patient self-report at 6 months. Secondary outcomes will include changes in HBA1c, weight, blood pressure, waist circumference, and levels of fasting lipids.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for study are adults (age ≥ 18) with type 2 diabetes who have a BMI 30-35, and are insured by Metroplus insurance, but otherwise meet NIH Consensus Criteria specifically (1) overweight for at least 5 years, (2) failure to lose weight with non-surgical means, (3) absence of medical or psychological contraindications, and (4) patient understanding of the procedure and its risks, and strong motivation to comply with the post-surgical regimen. Patients must have permission from their physician to participate in the study.

Exclusion Criteria:

Exclusions include being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks), participation in other obesity- or diabetes-related clinical trials, or diagnosis of cognitive dysfunction or significant psychiatric comorbidity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bariatric Clinic at Bellevue Hospital
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 6 months
  Within-patient change in insulin resistance after either bariatric surgery or initiation of intensive medical weight management, and remission of diabetes, (i.e., fasting glucose <126mg/dL and glucose <200mg/dL two hours after a standard 75g oral glucose load without the use of anti-hyperglycemic medications). Insulin resistance will be assessed at randomization and at 6 months with the homeostatic model assessment of insulin resistance (HOMA IR) based on insulin and fasting glucose, as well as oral glucose tolerance tests with area-under-the-curve (AUC) measurement for insulin values.

SECONDARY OUTCOMES:
Vitals status | 6 Months
  changes in HBA1c, weight, blood pressure, waist circumference, and levels of fasting lipids

CONTACTS AND LOCATIONS:
Locations (1):
- Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Parikh M, Chung M, Sheth S, McMacken M, Zahra T, Saunders JK, Ude-Welcome A, Dunn V, Ogedegbe G, Schmidt AM, Pachter HL. Randomized pilot trial of bariatric surgery versus intensive medical weight management on diabetes remission in type 2 diabetic patients who do NOT meet NIH criteria for surgery and the role of soluble RAGE as a novel biomarker of success. Ann Surg. 2014 Oct;260(4):617-22; discussion 622-4. doi: 10.1097/SLA.0000000000000919. PMID 25203878